CLINICAL TRIAL: NCT00601510
Title: A Phase I Study of Capecitabine, Cisplatin and Imatinib in Patients With Unresectable or Metastatic Gastric Cancer.
Brief Title: Imatinib, Capecitabine, and Cisplatin in Treating Patients With Unresectable or Metastatic Stomach Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000581134; KRDI-TUM-STI571; KRDI-TUM-GLIVEC-CSTI571BDE54; EU-20797; NOVARTIS-KRDI-TUM-STI571; EUDRACT-2006-005792-17
Record Dates: First submitted 2008-01-25; First posted 2008-01-28 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Gastric Cancer
Keywords: stage III gastric cancer; stage IV gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Cisplatin; Imatinib Mesylate

ARMS (1):
- Imatinib mesylate (Experimental): Imatinib mesylate 300mg/day(maximum dose will be 800 mg) on day -4, -3, -2, -1, 1, 2, 3 through d21 in combination with capecitabine 1250 mg/m2 twice daily (d1-d14) and iv cisplatin 60mg/m2
  Interventions: Drug: capecitabine; Drug: cisplatin; Drug: imatinib mesylate

INTERVENTIONS:
Drug: capecitabine
Drug: cisplatin
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Imatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as capecitabine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving imatinib together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of imatinib when given together with capecitabine and cisplatin in treating patients with unresectable or metastatic stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerable dose and assess the safety and tolerability of imatinib mesylate in combination with capecitabine and cisplatin in patients with unresectable or metastatic gastric cancer.

Secondary

* To assess the preliminary antitumor activity of this regimen in these patients.
* To assess the response with regard to the expression and/or mutation of the tyrosine kinase receptors PDGF-R and c-kit in gastric cancer.

OUTLINE: This is a dose-escalation study of imatinib mesylate.

Patients receive oral imatinib mesylate once daily on days -4 to 21 in course 1 and on days 1-21 in all subsequent courses, oral capecitabine twice daily on days 1-14, and cisplatin IV on day 1. Courses repeat every 3 weeks* for 12 months in the absence of disease progression or unacceptable toxicity.

NOTE: *First course is 25 days.

After completion of study therapy, patients are followed every 3 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed gastric cancer

  * Unresectable and/or metastatic disease
* Incurable with any conventional multimodality approach by interdisciplinary assessment of the local tumor board
* Immunohistochemical documentation of c-kit (CD117) and PDGF-R overexpression by tumor if obtainable (preferably on a tumor sample taken within 6 weeks of study entry)
* At least one evaluable site of disease according to RECIST criteria
* No known brain metastasis or CNS disorder that might alter study compliance or may worsen during or following therapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* WBC ≥ 3,000/μL
* ANC ≥ 2,000/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 9.0 g/dL
* Total bilirubin < 2 times upper limit of normal (ULN)
* SGOT and SGPT < 2.5 times ULN (5 times ULN if hepatic metastases present)
* Glomerular filtration rate ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for up to 3 months after completion of study treatment
* No known or documented hypersensitivity against fluoropyrimidines, tyrosine kinase inhibitors, cisplatin, other platinums, or their respective derivatives
* No gastrointestinal disorder that might affect the gastrointestinal absorption of capecitabine or imatinib mesylate or ability to swallow for the oral administration of capecitabine or imatinib mesylate
* At least 5 years since prior primary malignancy except if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or carcinoma in situ of the cervix
* No other concurrent malignant disease
* No NYHA class III-IV cardiac disease (i.e., congestive heart failure or myocardial infarction within the past 6 months)
* No severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection)
* No known neuropathy, impaired hearing, history of seizures, and/or psychiatric disorder that might alter study compliance or may worsen during or following therapy
* No documented dihydropyrimidine dehydrogenase deficiency
* No known chronic liver disease (i.e., chronic active hepatitis or cirrhosis)
* No known diagnosis of HIV infection or other serious uncontrolled infections
* No significant history of non-compliance to medical regimens or inability to grant reliable informed consent

PRIOR CONCURRENT THERAPY:

* No chemotherapy or investigational agents within the past 4 weeks (6 weeks for nitrosoureas or mitomycin C) unless the disease is rapidly progressing
* No prior radiotherapy to ≥ 25% of the bone marrow
* No major surgery within the past 2 weeks
* No concurrent warfarin or acetaminophen

  * Therapeutic anticoagulation using heparin or low-molecular weight heparin allowed
* No concurrent sorivudine or related substances
* No other concurrent anticancer agents, including chemotherapy and biologic agents
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-11; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Safety
Tolerability
Overall tumor response as assessed by RECIST

SECONDARY OUTCOMES:
Time to progression of disease
Overall survival
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Ebert, MD, Study Chair — Technical University of Munich
Locations (1):
- Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich, Germany

REFERENCES:
- [Derived] Mayr M, Becker K, Schulte N, Belle S, Hofheinz R, Krause A, Schmid RM, Rocken C, Ebert MP. Phase I study of imatinib, cisplatin and 5-fluoruracil or capecitabine in advanced esophageal and gastric adenocarcinoma. BMC Cancer. 2012 Dec 10;12:587. doi: 10.1186/1471-2407-12-587. PMID 23228190